CLINICAL TRIAL: NCT04831216
Title: Delivering Health: An Integrated Approach to Address Diabetes in the Context of Food Insecurity
Brief Title: Delivering Health: Addressing Diabetes and Food Insecurity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 260304
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Results first posted 2025-04-17 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-03

CONDITIONS: Food Insecurity; Diabetes Mellitus, Type 2
Keywords: Food insecurity; Type 2 diabetes mellitus; Nutrition; Food delivery
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: All participants will be assigned to a single intervention arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Type 2 Diabetes Appropriate Food Boxes + Diabetes Education (Experimental): All participants will be assigned to a single intervention arm. The intervention includes weekly delivery of type 2 diabetes-appropriate food boxes that include diabetes self-management education materials.
  Interventions: Behavioral: Type 2 Diabetes Appropriate Food Boxes + Diabetes Education

INTERVENTIONS:
Behavioral: Type 2 Diabetes Appropriate Food Boxes + Diabetes Education — All participants will be assigned to a single intervention arm. The intervention includes weekly delivery of type 2 diabetes-appropriate food boxes that include diabetes self-management education materials.

SUMMARY:
The goal of this study was to develop, implement, and evaluate the effectiveness of an intervention to use home-delivery of Type 2 diabetes (T2D)-appropriate food boxes with plain language adapted education materials to improve the nutritional health, physical activity, and health outcomes of low-income food insecure people with T2D in northwest Arkansas.

DETAILED DESCRIPTION:
Background and Rationale

Decades of increasing incidence of type 2 diabetes (T2D) present a multifaceted challenge to the health of a growing number of Americans, affecting their diets and how they live life. Approximately 30 million (~9%) of all people in the US have T2D, and this number is expected to continue to rise. At the same time, 15 million (11.8%) US households experience food insecurity, which is associated with risk for T2D and other chronic diseases. Both T2D and food insecurity are even more prevalent in Arkansas, with rates of T2D and food insecurity at 12.2% and 17.3%, respectively.

Approximately 46 million Americans per year turn to food pantries and related programs to help meet household nutritional needs. However, food pantries are not a long-term solution to improve health for food insecure people with T2D. Most food pantries do not provide food of sufficient dietary quality to support a healthy lifestyle.

Diabetes self-management education (DSME) is an approach with documented efficacy in helping people manage T2D. DSME supports informed decision-making, encourages goal setting and problem solving, and improves self-care behaviors. Recent studies have shown promise for DSME among food pantry clients with T2D. However, studies have suffered from problems with attendance and retention.

We designed a study to develop and evaluate the efficacy of a plain-language DSME curriculum to improve the nutritional health, physical activity, and health outcomes of low-income food insecure people with T2D. We home-delivered this curriculum along with T2D-appropriate healthy food boxes to mitigate difficulties associated with access to healthy food and attendance at DSME sessions outside of the home. We hypothesized that this approach will lead to improvements in participants' glycemic control, diet quality, and other outcomes.

Study Population Up to 110 study participants will be recruited from food pantries located in Benton and Washington Counties in northwest Arkansas.

Inclusion Criteria:

* 18 years of age or older
* Food insecure (confirmed with adapted 10-item screener)
* HbA1c levels of ≥7%

Exclusion Criteria:

* Conditions making it unlikely the participant will be able to follow the protocol, such as terminal illness, non-ambulatory, severe mental illness, severely impaired vision or hearing, eating disorder, or plans to move out of the geographic region
* Pregnant
* Only one adult per household will be enrolled

Study Design and Procedures For each participant, participation took place over 22 weeks (Weeks 1-4: Pre-intervention data collection; Weeks 5-16: Intervention; Weeks 17-22: Post-intervention data collection). Data collection took place at pre-intervention and post-intervention for each participant. At enrollment (i.e., pre-intervention) and one week after the 12th food box delivery (i.e. post-intervention), participants provided data on glycemic control (measured by HbA1c), physical activity, body mass index (BMI), T2D self-management behaviors, T2D knowledge, T2D self-efficacy, and food security. To enhance the study's significance in characterizing the diet patterns and fruit and vegetable consumption of low-income food insecure people with T2D, we collected extensive diet quality data measures pre-intervention and post-intervention.

Data Analysis To examine the intervention's effect on the primary outcomes of glycemic control as measured by HbA1c and diet quality as measured by Healthy Eating Index-2015 (HEI) scores, we used mixed effects regression models for repeated measures. These analyses focused on testing for a statistically significant difference between pre-intervention versus post-intervention measures. Analyses included relevant covariates such as sex or age.

ELIGIBILITY:
Inclusion Criteria

* 18 years of age or older
* Food insecure (confirmed with adapted 10-item screener)
* HbA1c levels of ≥7%

Exclusion Criteria

* Conditions making it unlikely the participant will be able to follow the protocol, such as terminal illness, non-ambulatory, severe mental illness, severely impaired vision or hearing, eating disorder, or plans to move out of the geographic region
* Pregnant
* Only one adult per household will be enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2021-08-24 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Krista N Langston, MBA, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences Northwest, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Type 2 Diabetes Appropriate Food Boxes + Diabetes Education
Started | 101
Completed | 69
Not Completed | 32
Not completed — Lost to Follow-up | 32

BASELINE CHARACTERISTICS:
Arm/Group | Type 2 Diabetes Appropriate Food Boxes + Diabetes Education
Number analyzed (Participants) | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 35
  Marshallese | 33
  White | 26
  Other | 7
Region of Enrollment [Number; unit: participants]
  United States | 101
Hemoglobin A1c (%) [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] | 9.87 (2.25)

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c (HbA1c), %
Description: A Siemens analyzer was utilized to measure HbA1c (%) via finger stick blood collection.
Time Frame: Baseline; immediate post-intervention (approx. 20 weeks)
Population: Analysis used all available data from participants.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Type 2 Diabetes Appropriate Food Boxes + Diabetes Education
Number analyzed (Participants) | 101
percentage of glycosylated hemoglobin
  Baseline | 9.87 (2.25)
  Post-intervention: number analyzed (Participants) | 69
  Post-intervention | 9.12 (2.04)
Statistical Analysis 1: Comparison: Type 2 Diabetes Appropriate Food Boxes + Diabetes Education; Linear mixed effects regression model for repeated measures used all available participant data. Analyses do not include imputed missing values; Test type: Other; p = 0.0107, Mixed Models Analysis — The p-value reflects results of analysis of change in HbA1c from baseline to post-intervention; Linear mixed effects regression model included time, age, household size, gender, race, education, and employment

2. Secondary Outcome: Diet Quality
Description: Total skin carotenoid level was measured using a Veggie Meter optical skin scanner using Raman Spectroscopy. The Veggie Meter produces a score from 0 to 800, with higher scores indicating greater skin carotenoid levels, which suggest a greater intake of fruits and vegetables.
Time Frame: Baseline; immediate post-intervention (approx. 20 weeks)
Population: Analysis used all available data from participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Type 2 Diabetes Appropriate Food Boxes + Diabetes Education
Number analyzed (Participants) | 100
units on a scale
  Baseline | 258.47 (105.69)
  Post-intervention: number analyzed (Participants) | 69
  Post-intervention | 261.65 (107.03)
Statistical Analysis 1: Comparison: Type 2 Diabetes Appropriate Food Boxes + Diabetes Education; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.7927, Mixed Models Analysis — The p-value reflects results of analysis of change in skin carotenoid levels from baseline to post-intervention; Linear mixed effects regression model included time, age, household size, gender, race, education, and employment

3. Secondary Outcome: Diet Quality (2)
Description: 24 hour dietary recalls was collected using the Nutrition Data System for Research (NDSR). NDSR was used to calculate Healthy Eating Index-2015 (HEI) scores. HEI is a metric used to assess the quality of a person's diet by comparing their food intake to the Dietary Guidelines for Americans, with a higher score indicating a diet that more closely aligns with recommended nutritional guidelines. HEI scores range from 0 to 100, where a higher score is better.
Time Frame: Baseline; immediate post-intervention (approx. 20 weeks)
Population: Analysis used all available data from participants.
Measure: Mean (Standard Deviation); unit: HEI score
Arm/Group | Type 2 Diabetes Appropriate Food Boxes + Diabetes Education
Number analyzed (Participants) | 81
HEI score
  Baseline | 59.98 (16.26)
  Post-intervention: number analyzed (Participants) | 62
  Post-intervention | 58.61 (13.14)
Statistical Analysis 1: Comparison: Type 2 Diabetes Appropriate Food Boxes + Diabetes Education; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.4651, Mixed Models Analysis — The p-value reflects results of analysis of change in HEI score from baseline to post-intervention; Linear mixed effects regression model included time, age, household size, gender, race, education, and employment

4. Secondary Outcome: Body Mass Index (BMI)
Description: Weight and height was used to compute a continuous measure of BMI (kilograms per square meter).
Time Frame: Baseline; immediate post-intervention (approx. 20 weeks)
Population: Analysis used all available data from participants.
Measure: Mean (Standard Deviation); unit: kilograms per square meter
Arm/Group | Type 2 Diabetes Appropriate Food Boxes + Diabetes Education
Number analyzed (Participants) | 101
kilograms per square meter
  Baseline | 33.42 (7.15)
  Post-intervention: number analyzed (Participants) | 68
  Post-intervention | 32.90 (5.76)
Statistical Analysis 1: Comparison: Type 2 Diabetes Appropriate Food Boxes + Diabetes Education; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.2439, Mixed Models Analysis — The p-value reflects results of analysis of change in BMI from baseline to post-intervention; Linear mixed effects regression model included time, age, household size, gender, race, education, and employment

5. Secondary Outcome: Chronic Diseases
Description: Self-report items from the Behavioral Risk Factor Surveillance System (BRFSS) survey assessed lifetime prevalence of chronic diseases.
Time Frame: Baseline; immediate post-intervention (approx. 20 weeks)
Population: There was a high degree of missingness on these items at baseline and post-intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Type 2 Diabetes Appropriate Food Boxes + Diabetes Education
Number analyzed (Participants) | 83
Participants
  Baseline: Reported one or more chronic diseases | 71
  Baseline: Did not report a chronic disease | 12
  Post-intervention: number analyzed (Participants) | 59
  Post-intervention: Reported one or more chronic diseases | 51
  Post-intervention: Did not report a chronic disease | 8

6. Secondary Outcome: Type 2 Diabetes Self-Management Self-Efficacy
Description: Self-efficacy for self-management of type 2 diabetes was assessed using the eight item Diabetes Self-Efficacy Scale (DSES). The DSES assesses confidence in a person's perceived capability to perform necessary type 2 diabetes self-care activities including, maintaining healthy diet, engaging in exercise, and performing blood sugar monitoring (0, Not at all confident to 10, Totally confident). The score for the scale is the mean of the eight items, producing a range of scores of 0-10, with higher scores indicating higher levels of confidence to perform diabetes self-management activities.
Time Frame: Baseline; immediate post-intervention (approx. 20 weeks)
Population: Analysis used all available data from participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Type 2 Diabetes Appropriate Food Boxes + Diabetes Education
Number analyzed (Participants) | 101
score on a scale
  Baseline | 6.88 (2.22)
  Post-intervention: number analyzed (Participants) | 69
  Post-intervention | 6.89 (2.23)
Statistical Analysis 1: Comparison: Type 2 Diabetes Appropriate Food Boxes + Diabetes Education; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.6794, Mixed Models Analysis — The p-value reflects results of analysis of change in DMSES scale score from baseline to post-intervention; Linear mixed effects regression model included time, age, household size, gender, race, education, and employment

7. Secondary Outcome: Oral Health
Description: Oral health was assessed by a single self-report item from the BRFSS, asking length of time since a dental cleaning ("Within the past year=1; Within the past 2 years=2; Within the past 5 years=3; 5 or more years ago=4; Never=5"). A lower score indicates a better outcome (more recent dental cleaning).
Time Frame: Baseline; immediate post-intervention (approx. 20 weeks)
Population: Analysis used all available data from participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Type 2 Diabetes Appropriate Food Boxes + Diabetes Education
Number analyzed (Participants) | 88
Participants
  Baseline: Within the past year | 36
  Baseline: Within the past 2 years | 17
  Baseline: Within the past 5 years | 10
  Baseline: 5 or more years ago | 9
  Baseline: Never | 16
  Post-intervention: number analyzed (Participants) | 62
  Post-intervention: Within the past year | 32
  Post-intervention: Within the past 2 years | 8
  Post-intervention: Within the past 5 years | 8
  Post-intervention: 5 or more years ago | 7
  Post-intervention: Never | 7
Statistical Analysis 1: Comparison: Type 2 Diabetes Appropriate Food Boxes + Diabetes Education; Cumulative logit mixed effects model (using PROC GLIMMIX) for repeated measures used all available participant data. This model is specifically designed for ordinal outcomes. Analyses do not include imputed missing values; Test type: Other; p = 0.1043, Mixed Models Analysis — The p-value reflects results of analysis of change in oral health behavior from baseline to post-intervention; Cumulative logit mixed effects model included time, age, household size, gender, race, education, and employment

8. Secondary Outcome: Type 2 Diabetes-related Distress
Description: Psychological distress related to type 2 diabetes was assessed using the Problem Areas in Diabetes 5-item scale (PAID-5) scale. The PAID-5 is used to assess the emotional distress related to living with type 2 diabetes, consisting of five questions that focus on feelings like fear, depression, worry about future complications, feeling overwhelmed by diabetes management, and coping with diabetes complications; essentially measuring the psychological impact of managing diabetes on a person's daily life (0, Not a problem to 4, Serious problem). The sum of the items produces a total score that ranges from 0-20, with lower scores indicating less distress.
Time Frame: Baseline; immediate post-intervention (approx. 20 weeks)
Population: Analysis used all available data from participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Type 2 Diabetes Appropriate Food Boxes + Diabetes Education
Number analyzed (Participants) | 101
score on a scale
  Baseline | 7.63 (6.17)
  Post-intervention: number analyzed (Participants) | 69
  Post-intervention | 4.28 (4.62)
Statistical Analysis 1: Comparison: Type 2 Diabetes Appropriate Food Boxes + Diabetes Education; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, Mixed Models Analysis — The p-value reflects results of analysis of change in PAID-5 scale score from baseline to post-intervention; Linear mixed effects regression model included time, age, household size, gender, race, education, and employment

9. Secondary Outcome: Food Security
Description: Food security was assessed using the Hunger Vital Sign two-question screening tool. Food security was not assessed at post-intervention, therefore no data can be reported for this measure.
Time Frame: Baseline
Population: Results are for baseline only. Food security was not assessed at post-intervention due to survey programming errors, therefore no outcome data can be reported for this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Type 2 Diabetes Appropriate Food Boxes + Diabetes Education
Number analyzed (Participants) | 101
Participants
  Baseline: Food insecure | 100
  Baseline: Food secure | 1
  Post-intervention: number analyzed (Participants) | 0

10. Secondary Outcome: Food Pantry Utilization
Description: Food pantry utilization was assessed through a single survey item adapted from Feeding America's Hunger in America survey. The item asked how many times the participant got food from a food pantry in the past 30 days.
Time Frame: Baseline; immediate post-intervention (approx. 20 weeks)
Population: Analysis used all available data from participants.
Measure: Mean (Standard Deviation); unit: times visited food pantry, past 30 days
Arm/Group | Type 2 Diabetes Appropriate Food Boxes + Diabetes Education
Number analyzed (Participants) | 101
times visited food pantry, past 30 days
  Baseline | 2.72 (2.65)
  Post-intervention: number analyzed (Participants) | 69
  Post-intervention | 2.48 (2.06)
Statistical Analysis 1: Comparison: Type 2 Diabetes Appropriate Food Boxes + Diabetes Education; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.5332, Mixed Models Analysis — The p-value reflects results of analysis of change in number of visits to food pantries in the past 30 days from baseline to post-intervention; Linear mixed effects regression model included time, age, household size, gender, race, education, and employment

11. Secondary Outcome: Medication Adherence
Description: Type 2 diabetes medication adherence was collected using responses to six items (0, No; 1, Yes) from the National Health Interview Survey (NHIS). The survey items assess how well individuals with diabetes adhered to their prescribed medication regimen, specifically by measuring whether they are taking medications correctly and refilling prescriptions as directed versus using non-adherence strategies to lower the cost of their medications (e.g., skipping doses, taking less medicine than prescribed, delaying filling prescriptions). Scores ranged from 0-6, with lower scores on the scale indicating a better outcome (e.g., better adherence to medication regimens).
Time Frame: Baseline; immediate post-intervention (approx. 20 weeks)
Population: Analysis used all available data from participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Type 2 Diabetes Appropriate Food Boxes + Diabetes Education
Number analyzed (Participants) | 101
score on a scale
  Baseline | 3.70 (2.10)
  Post-intervention: number analyzed (Participants) | 69
  Post-intervention | 3.07 (1.29)
Statistical Analysis 1: Comparison: Type 2 Diabetes Appropriate Food Boxes + Diabetes Education; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0468, Mixed Models Analysis — The p-value reflects results of analysis of change in ARMS-D scale scores from baseline to post-intervention; Linear mixed effects regression model included time, age, household size, gender, race, education, and employment

12. Secondary Outcome: Cooking Skills and Knowledge (1)
Description: Cooking skills and knowledge were assessed using two items. The first item asks "How confident do you feel being able to cook from raw or basic ingredients?" Response options include "Not confident at all; Somewhat confident; and Completely confident". Cooking skills and knowledge were not assessed at post-intervention, therefore no data can be reported for this measure.
Time Frame: Baseline
Population: Cooking skills and knowledge were not assessed at post-intervention due to survey programming errors, therefore no outcome data can be reported for this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Type 2 Diabetes Appropriate Food Boxes + Diabetes Education
Number analyzed (Participants) | 101
Participants
  Baseline: Completely confident | 92
  Baseline: Somewhat confident | 9
  Baseline: Not confident at all | 0
  Post-intervention: number analyzed (Participants) | 0

13. Secondary Outcome: Cooking Skills and Knowledge (2)
Description: Cooking skills and knowledge were assessed using two items. The second item asks "How confident do you feel about following a simple recipe?" Response options include "Not confident at all; Somewhat confident; and Completely confident". Cooking skills and knowledge were not assessed at post-intervention, therefore no data can be reported for this measure.
Time Frame: Baseline
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Type 2 Diabetes Appropriate Food Boxes + Diabetes Education
Number analyzed (Participants) | 101
Participants
  Baseline: Completely confident | 93
  Baseline: Somewhat confident | 8
  Baseline: Not confident at all | 0
  Post-intervention: number analyzed (Participants) | 0

14. Secondary Outcome: Type 2 Diabetes Self-Management Behaviors - General Diet
Description: The Summary of Diabetes Self-Care Activities (SDSCA) was used to assess self-management behaviors. The SDSCA is used to assess how well individuals with diabetes manage their condition by measuring the frequency (number of days) of their self-care practices like diet, exercise, blood glucose monitoring, and foot care over the past seven days.
  The General Diet subscale is 2 items assessing how many days participants adhered to a diet plan (0-7 days per week).
Time Frame: Baseline; immediate post-intervention (approx. 20 weeks)
Population: Analysis used all available data from participants.
Measure: Mean (Standard Deviation); unit: days per week
Arm/Group | Type 2 Diabetes Appropriate Food Boxes + Diabetes Education
Number analyzed (Participants) | 101
days per week
  Baseline | 2.32 (2.52)
  Post-intervention: number analyzed (Participants) | 69
  Post-intervention | 4.34 (2.17)
Statistical Analysis 1: Comparison: Type 2 Diabetes Appropriate Food Boxes + Diabetes Education; [analysis description as in outcome 1, analysis 1]; Test type: Other; p < 0.0001, Mixed Models Analysis — The p-value reflects results of analysis of change in days per week following general healthful diet from baseline to post-intervention; Linear mixed effects regression model included time, age, household size, gender, race, education, and employment

15. Secondary Outcome: Type 2 Diabetes Self-Management Behaviors - Specific Diet
Description: The Summary of Diabetes Self-Care Activities (SDSCA) was used to assess self-management behaviors. The SDSCA is used to assess how well individuals with diabetes manage their condition by measuring the frequency (number of days) of their self-care practices like diet, exercise, blood glucose monitoring, and foot care over the past seven days.
  The Specific Diet subscale is 2 items assessing how many days participants ate certain types of foods (0-7 days per week).
Time Frame: Baseline; immediate post-intervention (approx. 20 weeks)
Population: Analysis used all available data from participants.
Measure: Mean (Standard Deviation); unit: days per week
Arm/Group | Type 2 Diabetes Appropriate Food Boxes + Diabetes Education
Number analyzed (Participants) | 101
days per week
  Baseline | 3.83 (1.77)
  Post-intervention: number analyzed (Participants) | 69
  Post-intervention | 4.33 (1.64)
Statistical Analysis 1: Comparison: Type 2 Diabetes Appropriate Food Boxes + Diabetes Education; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0649, Mixed Models Analysis — The p-value reflects results of analysis of change in days per week following specific diet recommendations from baseline to post-intervention; Linear mixed effects regression model included time, age, household size, gender, race, education, and employment

16. Secondary Outcome: Type 2 Diabetes Self-Management Behaviors - Exercise
Description: The Summary of Diabetes Self-Care Activities (SDSCA) was used to assess self-management behaviors. The SDSCA is used to assess how well individuals with diabetes manage their condition by measuring the frequency (number of days) of their self-care practices like diet, exercise, blood glucose monitoring, and foot care over the past seven days.
  The Exercise subscale is 2 items assessing how many days participants engaged in exercise (0-7 days per week).
Time Frame: Baseline; immediate post-intervention (approx. 20 weeks)
Population: Analysis used all available data from participants.
Measure: Mean (Standard Deviation); unit: days per week
Arm/Group | Type 2 Diabetes Appropriate Food Boxes + Diabetes Education
Number analyzed (Participants) | 101
days per week
  Baseline | 2.07 (1.99)
  Post-intervention: number analyzed (Participants) | 69
  Post-intervention | 2.88 (2.30)
Statistical Analysis 1: Comparison: Type 2 Diabetes Appropriate Food Boxes + Diabetes Education; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0049, Mixed Models Analysis — The p-value reflects results of analysis of change in days per week engaging in exercise from baseline to post-intervention; Linear mixed effects regression model included time, age, household size, gender, race, education, and employment

17. Secondary Outcome: Type 2 Diabetes Self-Management Behaviors - Blood Glucose Testing
Description: The Summary of Diabetes Self-Care Activities (SDSCA) was used to assess self-management behaviors. The SDSCA is used to assess how well individuals with diabetes manage their condition by measuring the frequency (number of days) of their self-care practices like diet, exercise, blood glucose monitoring, and foot care over the past seven days.
  The Blood Glucose Testing subscale is 2 items assessing how many days participants tested their blood sugar (0-7 days per week).
Time Frame: Baseline; immediate post-intervention (approx. 20 weeks)
Population: Analysis used all available data from participants.
Measure: Mean (Standard Deviation); unit: days per week
Arm/Group | Type 2 Diabetes Appropriate Food Boxes + Diabetes Education
Number analyzed (Participants) | 101
days per week
  Baseline | 3.39 (2.93)
  Post-intervention: number analyzed (Participants) | 69
  Post-intervention | 4.39 (2.68)
Statistical Analysis 1: Comparison: Type 2 Diabetes Appropriate Food Boxes + Diabetes Education; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0086, Mixed Models Analysis — The p-value reflects results of analysis of change in days per week conducted blood glucose testing from baseline to post-intervention; Linear mixed effects regression model included time, age, household size, gender, race, education, and employment

18. Secondary Outcome: Type 2 Diabetes Self-Management Behaviors - Foot Care
Description: The Summary of Diabetes Self-Care Activities (SDSCA) was used to assess self-management behaviors. The SDSCA is used to assess how well individuals with diabetes manage their condition by measuring the frequency (number of days) of their self-care practices like diet, exercise, blood glucose monitoring, and foot care over the past seven days.
  The Foot Care subscale is 2 items assessing how many days participants performed a foot check and inspected the inside of their shoes (0-7 days per week).
Time Frame: Baseline; immediate post-intervention (approx. 20 weeks)
Population: Analysis used all available data from participants.
Measure: Mean (Standard Deviation); unit: days per week
Arm/Group | Type 2 Diabetes Appropriate Food Boxes + Diabetes Education
Number analyzed (Participants) | 101
days per week
  Baseline | 4.19 (2.83)
  Post-intervention: number analyzed (Participants) | 69
  Post-intervention | 4.72 (2.61)
Statistical Analysis 1: Comparison: Type 2 Diabetes Appropriate Food Boxes + Diabetes Education; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0243, Mixed Models Analysis — The p-value reflects results of analysis of change in days per week conducting food checks from baseline to post-intervention; Linear mixed effects regression model included time, age, household size, gender, race, education, and employment

19. Secondary Outcome: Type 2 Diabetes Self-Management Behaviors - Smoking
Description: The Summary of Diabetes Self-Care Activities (SDSCA) was used to assess self-management behaviors. The SDSCA is used to assess how well individuals with diabetes manage their condition by measuring the frequency (number of days) of their self-care practices like diet, exercise, blood glucose monitoring, and foot care over the past seven days. Smoking was assessed using a single yes/no item.
Time Frame: Baseline; immediate post-intervention (approx. 20 weeks)
Population: Analysis used all available data from participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Type 2 Diabetes Appropriate Food Boxes + Diabetes Education
Number analyzed (Participants) | 101
Participants
  Baseline: Yes | 16
  Baseline: No | 85
  Post-intervention: number analyzed (Participants) | 69
  Post-intervention: Yes | 11
  Post-intervention: No | 58
Statistical Analysis 1: Comparison: Type 2 Diabetes Appropriate Food Boxes + Diabetes Education; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.2861, Mixed Models Analysis — The p-value reflects results of analysis of change in smoking status (yes/no) from baseline to post-intervention; Linear mixed effects regression model included time, age, household size, gender, race, education, and employment

20. Secondary Outcome: Type 2 Diabetes Self-Management Behaviors - Medication Adherence
Description: The Summary of Diabetes Self-Care Activities (SDSCA) was used to assess self-management behaviors. The SDSCA is used to assess how well individuals with diabetes manage their condition by measuring the frequency (number of days) of their self-care practices like diet, exercise, blood glucose monitoring, and foot care over the past seven days.
  The Medication Adherence subscale is 2 items assessing how many days participants adhered to taking recommended diabetes medications (0-7 days per week).
Time Frame: Baseline; immediate post-intervention (approx. 20 weeks)
Population: Analysis used all available data from participants.
Measure: Mean (Standard Deviation); unit: days per week
Arm/Group | Type 2 Diabetes Appropriate Food Boxes + Diabetes Education
Number analyzed (Participants) | 101
days per week
  Baseline | 2.43 (3.23)
  Post-intervention: number analyzed (Participants) | 68
  Post-intervention | 2.26 (3.23)
Statistical Analysis 1: Comparison: Type 2 Diabetes Appropriate Food Boxes + Diabetes Education; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.9933, Mixed Models Analysis — The p-value reflects results of analysis of change in days per week adhering to prescribed medications from baseline to post-intervention; Linear mixed effects regression model included time, age, household size, gender, race, education, and employment

ADVERSE EVENTS:
Time Frame: From enrollment to approximately 20 weeks post-intervention
Description: Study staff assessed adverse events via regular contact with participants throughout the duration of the study.
Arm/Group | Type 2 Diabetes Appropriate Food Boxes + Diabetes Education
All-Cause Mortality (participants affected / at risk) | 0/101
Serious Adverse Events (participants affected / at risk) | 0/101
Other Adverse Events (participants affected / at risk) | 0/101

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/16/NCT04831216/Prot_SAP_000.pdf
  • Informed Consent Form (2023-02-08): https://cdn.clinicaltrials.gov/large-docs/16/NCT04831216/ICF_001.pdf